CLINICAL TRIAL: NCT01097018
Title: A Phase III Randomized Study to Assess the Efficacy and Safety of Perifosine Plus Capecitabine Versus Placebo Plus Capecitabine in Patients With Refractory Advanced Colorectal Cancer
Brief Title: Perifosine Plus Capecitabine Versus Placebo Plus Capecitabine in Patients With Refractory Advanced Colorectal Cancer
Acronym: X-PECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol 343
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; perifosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perifosine + Capecitabine (Active Comparator): Perifosine 1 tablet daily + Capecitabine BID days 1 - 14 every 21 days
  Interventions: Drug: Capecitabine; Drug: Perifosine
- Placebo + Capecitabine (Placebo Comparator): Placebo 1 tablet daily + Capecitabine BID days 1 - 14 every 21 days
  Interventions: Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m2 BID/ Days 1-14
Drug: Perifosine — 50 mg daily x 21 days
  Arms: Perifosine + Capecitabine
Drug: Placebo — 1 pill daily x 21 days
  Arms: Placebo + Capecitabine

SUMMARY:
The trial will compare the overall survival of perifosine plus capecitabine to placebo plus capecitabine in patients with refractory advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have failed available therapy for the treatment of advanced colorectal cancer, including fluoropyrimidine, irinotecan, oxaliplatin, bevacizumab and for K-ras wild-type (WT) patients, anti-EGFR antibody (cetuximab or panitumumab) containing therapies.
* For oxaliplatin-based therapy, failure of therapy will also include patients who had oxaliplatin discontinued secondary to toxicity.
* No prior exposure to capecitabine in the metastatic colorectal cancer setting, except limited-course radiosensitizing capecitabine
* Patients must have at least one measurable lesion by RECIST criteria

Exclusion Criteria:

* Patients with known dipyrimidine dehydrogenase (DPD) deficiency or prior severe reaction to 5-FU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Monthly

SECONDARY OUTCOMES:
Progression-free Survival | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (62):
- United States (62):
  - Alhambra, California
  - Bakersfield, California
  - La Verne, California
  - Long Beach, California
  - Los Angeles, California
  - Northridge, California
  - Redondo Beach, California
  - Santa Barbara, California
  - Santa Maria, California
  - Denver, Colorado
  - Grand Junction, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Stamford, Connecticut
  - Waterbury, Connecticut
  - Fort Myers, Florida
  - Hollywood, Florida
  - Pembroke Pines, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Lawrenceville, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Harvey, Illinois
  - Park Ridge, Illinois
  - South Bend, Indiana
  - Terre Haute, Indiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Lansing, Michigan
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Armonk, New York
  - Great Neck, New York
  - New Hyde Park, New York
  - New York, New York
  - Charlotte, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - TN Oncology, Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Midland, Texas
  - Tyler, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- [Result] Results of the X-PECT study: A phase III randomized double-blind, placebo-controlled study of perifosine plus capecitabine (P-CAP) versus placebo plus capecitabine (CAP) in patients (pts) with refractory metastatic colorectal cancer (mCRC). https://meetinglibrary.asco.org/content/98646-114 Abstract Number:LBA3501